CLINICAL TRIAL: NCT01011270
Title: Rehabilitation of Dynamic Muscle, Back Pain and Postural Balance of Industrial Operators
Brief Title: Rehabilitation of Dynamic Muscle, Back Pain and Postural Balance
Acronym: RDM
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universidade Camilo Castelo Branco (Other)
Responsible Party: Francisco Miguel Pinto, Universidade Castelo Branco
Other Study IDs: RDM - 0012009; RDM0012009UCB (Other Grant/Funding Number: UNIVERSIDADE CASTELO BRANCO)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Low Back Pain
Keywords: Back pain; postural balance; RDM; industrial operators
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Back pain: The aim of this study was to investigate the effect of rehabilitation of the dynamic ;(RDM) in balance and balance of industrial operators. The sample consisted of industrial operators, individuals with low back pain, referred to the industry of Physical Therapy
- Balance: the treatment with RDM reflected in significant improvement in back pain and postural balance of industrial operators.

SUMMARY:
Workers in the various branches of the investigators industrial society can be considered as a group susceptible to risks due to the nature of its activities related to the intense demands of their work units with varying degrees of physical overload. Among the risk factors involved in postural genesis of occupational low back pain is work in uncomfortable positions, such as maintenance of static postures for long periods of time and frequent implementation of flexion, extension and trunk rotation.The association between body instability (lack of postural balance) and back pain is seen with some frequency, especially in working groups.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of rehabilitation of the dynamic muscle (RDM®) in back pain and postural balance of industrial operators. The sample consisted of industrial operators, individuals with low back pain, referred to the industry of Physical Therapy. After the screening criteria of inclusion and exclusion, 82 individuals were randomly selected and divided at random in: experimental group (GE, n = 41, age = 41 ± 4 years, body mass index (IMC) = 26.46 ± 3 , 25) and control group (CG, n = 42, age = 42 ± 5 years, IMC = 26.47 ± 3.34).

The GE was part of treatment with RDM. The CG was composed of individuals who did not participate in any physical therapy treatment during the search. The procedures used for evaluation were: back pain (Borg scale) and postural balance (pedana stabilometric and posturométrica). The process of intervention by the RDM had a duration of 20 minutes, frequency of twice a week and was extended for 12 weeks, and the systematic treatment performed on 4 occasions.

ELIGIBILITY:
Inclusion Criteria:

* FCC officials with medical indication of low back pain to perform physical therapy or medical

Exclusion Criteria:

* The investigators excluded patients who were doing treatment with medication and who reported worsening of the crisis period.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample consisted of industrial operators, individuals with low back pain, referred to the industry of Physical Therapy. After the screening criteria of inclusion and exclusion, 82 individuals
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
In intra-group comparison, the paired t test or Wilcoxon showed, respectively, a significant improvement (p <0.05) in the variables back pain (p = 0.0001) and postural balance (p = 0.0001) in GE. | three months

SECONDARY OUTCOMES:
Kruskal Wallis test followed by the confidence interval (CI) showed significant improvements in favor of GE's post-test compared to post-test of the GC (back pain: CI: -115.58 / -48.66; postural balance: CI: -68.81 / -1.89). | three months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Miguel, 3 Grau, Principal Investigator — Castelo Branco
Locations (1):
- Francisco Miguel Pinto, Rio de Janeiro, Rio de Janeiro, Brazil